CLINICAL TRIAL: NCT00818207
Title: A Pragmatic, Randomized, Controlled Study Evaluating The Impact Of Access To Smoking Cessation Treatment Reimbursement On The Proportion Of Successful Quitters In A Canadian Population Of Smokers Motivated To Quit
Brief Title: Impact Of Smoking Cessation Treatment Reimbursement On The Quit Rates In Smokers Motivated To Quit
Acronym: ACCESSATION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A3051116
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-02

CONDITIONS: Smoking Cessation; Insurance Coverage
Keywords: Smoking cessation; quit rates; reimbursement; drug coverage; effectiveness; cost-effectiveness; health policy; drug utilization; adherence; urine cotinine.
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Smoking Cessation Treatment Coverage (100%) (Other): A subject randomized to the intervention group will be eligible for smoking cessation treatment (SCT) reimbursement during the 26-week period following the randomization.
  Interventions: Other: Full Smoking Cessation Treatment Coverage (100%)
- No Smoking Cessation Treatment Coverage (0%) (Other): Subjects in the control group choosing to quit using an SCT method will not be eligible for smoking cessation treatment (SCT) reimbursement and, thus, will have to purchase their treatment out of pocket.
  Interventions: Other: No Smoking Cessation Treatment Coverage (0%)

INTERVENTIONS:
Other: Full Smoking Cessation Treatment Coverage (100%) — This is a pragmatic study in which the intervention is a health policy (SCT reimbursement). Champix (varenicline), Zyban (bupropion) and NRTs (nicotine replacement therapies; patches, gums) are SCT eligible for reimbursement. Prescriptions will be issued as per the most recent version of the Product Monograph of the prescribed SCT or equivalent.
  Arms: Full Smoking Cessation Treatment Coverage (100%)
Other: No Smoking Cessation Treatment Coverage (0%) — None of the subjects recruited in the study have access to SCT reimbursement in real-life. As such, subjects randomized to the control group represent lack of SCT coverage in real-life and are considered to receive standard of care for smoking cessation.
  Arms: No Smoking Cessation Treatment Coverage (0%)

SUMMARY:
This study is based on the hypothesis that access to smoking cessation treatment (SCT) reimbursement may significantly increase the number of successful quitters in a population of smokers motivated to quit by: 1) increasing the use of SCTs in quit attempts, and 2) by improving subject adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Daily smokers (10 cigarettes per day or more);
* Smokers motivated to make a quit attempt within the next 14 days;
* Potential subjects must be outpatients;
* A subject must have a stable mental and physical medical condition (as per investigator's judgment).

Exclusion Criteria:

* A subject currently eligible for smoking cessation treatment (SCT) reimbursement, whether from a public or a private drug insurance;
* A subject with an unknown drug insurance status;
* A subject living in a household where there is someone already recruited in the study;
* A subject with an unfilled SCT prescription issued within the past three months or with an unused SCT product;
* A subject with a life-threatening illness (ie, known or suspected cancer or other disease with a life expectancy of less than one year).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1380 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- Canada (34):
  - Pfizer Investigational Site, Burnaby, British Columbia
  - Pfizer Investigational Site, Chilliwack, British Columbia
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Kamloops, British Columbia
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Langley, British Columbia
  - Pfizer Investigational Site, North Vancouver, British Columbia
  - Pfizer Investigational Site, Penticton, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Bay Roberts, Newfoundland and Labrador
  - Pfizer Investigational Site, Paradise, Newfoundland and Labrador
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Sydney, Nova Scotia
  - Pfizer Investigational Site, Windsor, Nova Scotia
  - Pfizer Investigational Site, Aylmer, Ontario
  - Pfizer Investigational Site, Bolton, Ontario
  - Pfizer Investigational Site, Collingwood, Ontario
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Stayner, Ontario
  - Pfizer Investigational Site, Strathroy, Ontario
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Woodstock, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, Montague, Prince Edward Island
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Selby P, Brosky G, Oh P, Raymond V, Arteaga C, Ranger S. A pragmatic, randomized, controlled study evaluating the impact of access to smoking cessation pharmacotherapy coverage on the proportion of successful quitters in a Canadian population of smokers motivated to quit (ACCESSATION). BMC Public Health. 2014 May 7;14:433. doi: 10.1186/1471-2458-14-433. PMID 24885542
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051116&StudyName=Impact%20Of%20Smoking%20Cessation%20Treatment%20Reimbursement%20On%20The%20Quit%20Rates%20In%20Smokers%20Motivated%20To%20Quit

RESULTS

PARTICIPANT FLOW:
Groups:
- Reimbursement for Smoking Cessation Therapy (SCT): Participants used SCT of their choice, either pharmacological or non-pharmacological, or they could have chosen to use no SCT during the study. Participants in this group were fully reimbursed for the SCT used during the 26-week period following randomization.
- No Reimbursement for SCT: Participants used SCT of their choice, either pharmacological or non-pharmacological, or they could have chosen to use no SCT during the study. Participants in this group received no reimbursement for the SCT used during the 26-week period following randomization and had to pay for therapies out-of-pocket.
Period: Overall Study
Arm/Group | Reimbursement for Smoking Cessation Therapy (SCT) | No Reimbursement for SCT
Started | 696 | 684
Completed | 474 | 417
Not Completed | 222 | 267
Not completed — Adverse Event | 6 | 0
Not completed — Lost to Follow-up | 160 | 146
Not completed — Multiple reasons | 11 | 12
Not completed — Withdrawal by Subject | 42 | 104
Not completed — Death | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reimbursement for Smoking Cessation Therapy (SCT) | No Reimbursement for SCT | Total
Number analyzed (Participants) | 696 | 684 | 1380
Age Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (12.3) | 46.7 (12.3) | 46.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 342 | 347 | 689
  Male | 354 | 337 | 691

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 7-Day Point Prevalence (PP) of Abstinence
Description: Percentage of participants who self-reported tobacco abstinence for the previous 7 days (7-day PP) with a negative response to the following questions: "Have you smoked any cigarettes (even a puff) in the last 7 days?" and "Have you used any nicotine-containing product (such as chew, snuff, pipe, cigar) other than a Nicotine Replacement Therapy (NRT) (smoking cessation treatment [SCT]) in the last 7 days?"
Time Frame: Week 26
Population: Intent to Treat (ITT) Population: all randomized participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Reimbursement for Smoking Cessation Therapy (SCT) | No Reimbursement for SCT
Number analyzed (Participants) | 696 | 684
Percentage of Participants | 20.8 | 13.9
Statistical Analysis 1: Comparison: Reimbursement for Smoking Cessation Therapy (SCT) vs No Reimbursement for SCT; Odds ratios and p-values were obtained from a logistic regression model including the main effects of intervention and pooled center; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.23 to 2.18]

2. Secondary Outcome: Percentage of Participants With Biochemically Confirmed 7-Day PP Abstinence From Tobacco
Description: PP tobacco abstinence was adjudicated if the following conditions were met:(a) self-reported tobacco abstinence for the previous 7 days with a negative response to the questions "Have you smoked any cigarettes (even a puff) in the last 7 days?" and "Have you used any nicotine-containing product (such as chew, snuff, pipe, cigar) other than an NRT (SCT) in the last 7 days?" confirmed by negative urine cotinine test results (defined as cotinine levels less than [<]200 nanograms per milliliter [ng/mL]).
Time Frame: Week 26
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Reimbursement for Smoking Cessation Therapy (SCT) | No Reimbursement for SCT
Number analyzed (Participants) | 696 | 684
Percentage of Participants | 15.7 | 10.1
Statistical Analysis 1: Comparison: Reimbursement for Smoking Cessation Therapy (SCT) vs No Reimbursement for SCT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.21 to 2.33]

3. Secondary Outcome: Percentage of Participants With Continuous Abstinence (CA) at Weeks 26, 39, and 52
Description: CA from smoking was adjudicated if the following conditions were met:(a) self-reported continuous tobacco abstinence during the defined time point with a negative response to the questions "Have you smoked any cigarettes (even a puff) since the last contact/visit?" at every visit from Week 26 through Week 52 (Weeks 26, 39, and 52) and "Have you used any nicotine-containing product (such as chew, snuff, pipe, cigar) other than an NRT (SCT) since the last contact/visit?" and (b) urine cotinine test results were neither positive (greater than or equal to [≥]200 ng/mL) nor missing.
Time Frame: Week 26, Week 39, and Week 52
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Reimbursement for Smoking Cessation Therapy (SCT) | No Reimbursement for SCT
Number analyzed (Participants) | 696 | 684
Percentage of Participants
  Week 26 | 15.7 | 10.1
  Week 39 | 7.8 | 6.3
  Week 52 | 6.6 | 5.6
Statistical Analysis 1: Comparison: Reimbursement for Smoking Cessation Therapy (SCT) vs No Reimbursement for SCT; Week 39 odds ratios and p-values were obtained from a logistic regression model including the main effects of intervention and pooled center; Test type: Superiority or Other; p = 0.2979, Regression, Logistic — p-value was not adjusted for multiple comparisons; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.82 to 1.90]
Statistical Analysis 2: Comparison: Reimbursement for Smoking Cessation Therapy (SCT) vs No Reimbursement for SCT; Week 52 odds ratios and p-values were obtained from a logistic regression model including the main effects of intervention and pooled center; Test type: Superiority or Other; p = 0.4388, Regression, Logistic — p-value was not adjusted for multiple comparisons; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.76 to 1.87]

4. Secondary Outcome: Percentage of Participants With 7-Day PP of Abstinence at Week 13
Description: PP tobacco abstinence was adjudicated if the participant self-reported tobacco abstinence for the previous 7 days with a negative response to the following questions: "Have you smoked any cigarettes (even a puff) in the last 7 days?" and "Have you used any nicotine-containing product (such as chew, snuff, pipe, cigar) other than a NRT (SCT) in the last 7 days?"
Time Frame: Week 13
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Reimbursement for Smoking Cessation Therapy (SCT) | No Reimbursement for SCT
Number analyzed (Participants) | 696 | 684
Percentage of Participants | 34.1 | 23.7
Statistical Analysis 1: Comparison: Reimbursement for Smoking Cessation Therapy (SCT) vs No Reimbursement for SCT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value was not adjusted for multiple comparisons; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.35 to 2.20]

5. Secondary Outcome: Percentage of Participants With Long Term Quit Rate (LTQR) Through Weeks 26 to 52
Description: LTQR was adjudicated if the following conditions were met: the participant self-reported tobacco abstinence for the previous 7 days with a negative response to the following questions: "Have you smoked any cigarettes (even a puff) in the last 7 days?" and "Have you used any nicotine-containing product (such as chew, snuff, pipe, cigar) other than a NRT (SCT) in the last 7 days?" and had no more than 6 cumulative days of using nicotine containing products from Weeks 26 to 52
Time Frame: Week 26 to Week 52
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Reimbursement for Smoking Cessation Therapy (SCT) | No Reimbursement for SCT
Number analyzed (Participants) | 696 | 684
Percentage of Participants
  Week 26 | 20.8 | 13.9
  Week 30 | 19.7 | 12.6
  Week 34 | 17.4 | 12.3
  Week 39 | 14.9 | 11.3
  Week 44 | 13.7 | 11.0
  Week 48 | 12.5 | 10.8
  Week 52 | 11.2 | 9.9
Statistical Analysis 1: Comparison: Reimbursement for Smoking Cessation Therapy (SCT) vs No Reimbursement for SCT; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.4551, Regression, Logistic — p-value was not adjusted for multiple comparisons; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.81 to 1.62]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Reimbursement for Smoking Cessation Therapy (SCT) | No Reimbursement for SCT
Serious Adverse Events (participants affected / at risk) | 35/696 | 25/684
Other Adverse Events (participants affected / at risk) | 335/696 | 246/684
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reimbursement for Smoking Cessation Therapy (SCT) (N=696) | No Reimbursement for SCT (N=684)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Post procedural infection (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 1
Dissociative identity disorder (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0
Violence-related symptom (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reimbursement for Smoking Cessation Therapy (SCT) (N=696) | No Reimbursement for SCT (N=684)
Constipation (Gastrointestinal disorders) | 21 | 19
Diarrhoea (Gastrointestinal disorders) | 11 | 18
Dyspepsia (Gastrointestinal disorders) | 14 | 7
Nausea (Gastrointestinal disorders) | 107 | 50
Vomiting (Gastrointestinal disorders) | 17 | 13
Fatigue (General disorders) | 15 | 11
Irritability (General disorders) | 17 | 5
Bronchitis (Infections and infestations) | 21 | 22
Influenza (Infections and infestations) | 18 | 18
Nasopharyngitis (Infections and infestations) | 18 | 12
Sinusitis (Infections and infestations) | 17 | 12
Upper respiratory tract infection (Infections and infestations) | 30 | 24
Fall (Injury, poisoning and procedural complications) | 10 | 14
Weight increased (Investigations) | 16 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 17
Headache (Nervous system disorders) | 45 | 27
Abnormal dreams (Psychiatric disorders) | 55 | 18
Anxiety (Psychiatric disorders) | 28 | 17
Depression (Psychiatric disorders) | 30 | 26
Insomnia (Psychiatric disorders) | 41 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Rash (Skin and subcutaneous tissue disorders) | 16 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.